CLINICAL TRIAL: NCT03515382
Title: A Phase I, Open-Label, Randomized, Drug-Drug Interaction Study to Evaluate the Effect of Itraconazole and Voriconazole on the Single-Dose Pharmacokinetics of GLPG1690 in Healthy Male Subjects
Brief Title: A Study in Healthy Male Volunteers to Look at How the Test Medicine GLPG1690 is Taken up by the Body When Doses of Itraconazole and Voriconazole Are Given to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG1690-CL-106; 2017-004357-16 (EudraCT Number)
Record Dates: First submitted 2018-04-20; First posted 2018-05-03 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG1690; Itraconazole; Voriconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): single dose GLPG1690.
  Interventions: Drug: GLPG1690
- Treatment B (Experimental): Single dose itraconazole + single dose GLPG1690.
  Interventions: Drug: GLPG1690; Drug: Itraconazole
- Treatment C (Experimental): Single dose voriconazole + single dose GLPG1690.
  Interventions: Drug: GLPG1690; Drug: Voriconazole

INTERVENTIONS:
Drug: GLPG1690 — A single oral dose of GLPG1690.
Drug: Itraconazole — A single oral dose of itraconazole.
  Arms: Treatment B
Drug: Voriconazole — A single oral dose of voriconazole.
  Arms: Treatment C

SUMMARY:
The sponsor wants to investigate how well the test medicine is taken up by the body when given alongside two other already approved medicines. This kind of study is known as a drug-drug interaction study. In this case the other medicines are itraconazole and voriconazole.

The sponsor will also look at the safety and tolerability of the test medicine when taken alone, and when taken with the approved medicines.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed and dated informed consent form (ICF) as approved by the Independent Ethics Committee (IEC), prior to any screening evaluations.
* Male subject between 18-55 years of age (extremes included) on the day of signing the ICF.
* Body mass index (BMI) between 18.0-32.0 kg/m², inclusive, with body weight at least 50 kg.
* Judged by the investigator to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory results.
* Non-smoker, defined as an individual who has abstained from smoking (or the use of e-cigarettes or nicotine containing products) from at least 1 year prior to screening. A breath carbon monoxide reading of less than or equal to 10 ppm at screening and admission.
* Negative urine drug screen (at a minimum: amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone, and tricyclic antidepressants) and alcohol breath test at screening and admission.
* Negative serology for human immunodeficiency virus (HIV) type 1 or 2, hepatitis B virus surface antigen (HBs-Ag) or hepatitis C virus antibody (HCV-Ab), or any history of hepatitis from any cause, with the exception of hepatitis A at screening.
* Subject must agree to use highly effective contraceptive measures as and must be able and willing to comply with the other prohibitions and restrictions as described in the protocol.

Exclusion Criteria:

* History of serious allergic reaction to any drug as determined by the investigator (e.g. anaphylaxis requiring hospitalization) and/or known sensitivity to study drug or the excipients.
* Use of strong inhibitors and/or inducers of CYP3A4/5 and/or P-gp, including consumption of herbal medications (e.g. St. John's Wort) and grapefruit/grapefruit products within 7 days prior to the first study drug administration.
* Contra-indication for the use of itraconazole or voriconazole as described in the package insert.
* Abnormal liver function test, defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total bilirubin and/or gamma-glutamyl transferase (GGT) > 1.5 x upper limit of normal (ULN). Retesting is allowed once. Subjects with documented Gilbert's syndrome are eligible for inclusion in the study.
* History of malignancy within the past 5 years (except for basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
* Clinically relevant abnormalities detected on ECG regarding either rhythm, rate or conduction (e.g. QT interval corrected for the heart rate using Fridericia's formula [QTcF] ≥450 ms, or a known long QT syndrome). A first degree heart block or sinus arrhythmia is not considered as a significant abnormality.
* Clinically relevant abnormal vital signs and/or abnormalities detected during physical examination.
* Per judgment of the investigator, substantial blood loss (including blood donation), or a transfusion of any blood product within 8 weeks prior to the first study drug administration.
* Any condition or circumstances that, in the opinion of the investigator, could make a subject unlikely or unable to complete the study or comply with study procedures and requirements.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration of GLPG1690 (Cmax). | At various time points between Day 1 pre-dose and Day 5
  To investigate the effect of a single oral dose of itraconazole or voriconazole on the single-dose pharmacokinetics of GLPG1690 in healthy male subjects.
Area under the plasma concentration-time curve from time zero to infinity of GLPG1690 (AUC0-∞). | At various time points between Day 1 pre-dose and Day 5
  To investigate the effect of a single oral dose of itraconazole or voriconazole on the single-dose pharmacokinetics of GLPG1690 in healthy male subjects.
Apparent terminal half-life of GLPG1690 (t1/2,λz). | At various time points between Day 1 pre-dose and Day 5
  To investigate the effect of a single oral dose of itraconazole or voriconazole on the single-dose pharmacokinetics of GLPG1690 in healthy male subjects.

SECONDARY OUTCOMES:
Number of incidents of TEAEs. | Between screening and 10 days after the last dose
  To assess safety and tolerability of GLPG1690.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Brearley, BM, MRCP, MFPM, Study Director — Galapagos NV
Locations (1):
- Quotient Sciences Limited, Ruddington, United Kingdom